CLINICAL TRIAL: NCT03266926
Title: Does the Use of Bupivacaine Soaked Vaginal Packing Following Vaginal Surgery Decrease Postoperative Pain?
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: SBK Vaginal Pack Study
Record Dates: First submitted 2017-08-24; First posted 2017-08-30 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Pelvic Organ Prolapse; Postoperative Pain
MeSH Terms: conditions — Pelvic Organ Prolapse; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Postoperative Patients with premarin: Patients who undergo vaginal surgery at Sunnybrook Health Sciences Centre (SHSC) who require vaginal packing postoperatively and receive premarin vaginal cream coated packing.
  Interventions: Drug: Premarin Vaginal cream
- Postoperative Patients with bupivacaine: Patients who undergo vaginal surgery at Patients who undergo vaginal surgery (SHSC) who require vaginal packing postoperatively and receive bupivacaine soaked packing.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — 0.25% Bupivacaine with epinephrine will be applied to vaginal packing that is placed post vaginal reconstruction surgery.
  Other Names: Marcaine
  Groups: Postoperative Patients with bupivacaine
Drug: Premarin Vaginal cream — A Premarin vaginal cream will be used to coat the vaginal pack, prior to insertion in patients post vaginal reconstruction surgery.
  Other Names: estrogen vaginal cream
  Groups: Postoperative Patients with premarin

SUMMARY:
In current practice, packing in the vagina overnight after vaginal surgery is typically used to prevent post-surgical vaginal bleeding. The vaginal packing is usually coated with either estrogen cream or bupivacaine at the investigators' hospital . There are reports in the literature that show nasal packing soaked with local anesthetic after nasal sinus surgery reduces post-surgical pain. To date, no studies have evaluated local anesthetic soaked vaginal packing after vaginal surgery and if this is associated with a reduction in post-surgical pain scores.

The investigators seek to investigate if vaginal packing soaked with a local anesthetic reduces post-operative pain while providing the necessary action of minimizing potential post-surgical bleeding.

DETAILED DESCRIPTION:
This is a prospective cohort, single centre, single-blinded study looking at a population of women post vaginal surgery with vaginal packing that is either coated with estrogen cream or 0.25% Bupivacaine + epinephrine (local anesthetic). Patients who have booked vaginal surgery for prolapse repair will be invited to participate in this study. A document describing the study will be provided for reading and will include the consent for the study. At the end of surgery, a vaginal pack is placed to decrease potential bleeding post surgery. At this time, patients will receive either vaginal packing with estrogen, or, the vaginal packing with 0.25% bupivacaine + epinephrine, according to physician preference. Patients and the nurses caring for them post surgery will be blinded as to which group the patient has been assigned to. The nurses in the recovery room and post operative ward will ask patients post surgery the day of surgery, (POD#0, two and six hours post OR) and POD#1 to rate the patients' surgical pain with a standardized, validated VAS pain score. Secondary outcomes will be recorded: the amount of analgesics used in hospital after surgery, intra-operative blood loss, post operative hemoglobin, the number of days until the patient is able to void, the amount of analgesics used at home after surgery (patients will be asked to keep a record of the total number of oral analgesic pain tablets used and on which day post surgery they stopped using pain medications) and other post surgical complications. Data will be stored in a secure, password protected desktop on site. Each patient will be assigned a unique number which can be traced back to a master file which will include patient identifiers (name, MRN, DOB). Data will be analyzed with the appropriate statistical tests. There are no additional tests or visits for patients. Patient study assignment will be disclosed to them at the 6 week routine post surgical examination/assessment visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 4 attending physicians (urogynecologists) of Sunnybrook Health Sciences Centre planning to undergo a vaginal hysterectomy and/or vaginal reconstructive surgery for pelvic organ prolapse.
* Subjects aged 18 years and older and able to provide informed consent

Exclusion Criteria:

* Any patient undergoing abdominal prolapse repair or no vaginal repairs
* Patients undergoing vaginal obliterative procedures
* Patients with a known allergy or adverse reaction to Bupivacaine or contraindication to Premarin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants are eligible if they are undergoing vaginal reconstructive surgery.
Study Population: Women undergoing vaginal reconstructive surgery at Sunnybrook Health Sciences Centre.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | The outcome measure will be assessed six hours postoperative
  Primary outcome is postoperative pain score 6 hours post surgery on POD#0

SECONDARY OUTCOMES:
Intraoperative Blood Loss | One time measurement, intra-operative
  Estimate by the surgeon regarding total blood loss
Postoperative Hemoglobin | Morning of postoperative day one
  Measure of hemoglobin on the morning of postoperative day one
Analgesic Use In Hospital | From when surgery ends to time of discharge from hospital post operative day 1
  Compilation of total dose of Tylenol, anti-inflammatory, and narcotic use postoperatively
Post-operative per vaginal blood loss | From when surgery ends to time of discharge from hospital post operative day 1
  As subjectively described by RN in chart
Trial of Void | Up to six weeks postoperative
  Number of days required by the patient to pass a trial of void
Analgesic Use Postoperative | Up to six weeks postoperative
  Compilation of total dose of Tylenol, anti-inflammatory, and narcotic use from date of discharge to six week follow up
Visual Analog Scale (VAS) | The outcome measure will be assessed two hours postoperative
  postoperative pain score 2 hours post surgery on POD#0
Visual Analog Scale (VAS) | The outcome measure will be assessed on the morning of postoperative day one.
  postoperative pain score on the morning of postoperative day one

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Lee, MD, Principal Investigator — Sunnybrook Health Sciences Centre, University of Toronto
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdullah B, Khong SY, Tan PC. Oestrogen-soaked vaginal packing for decubitus ulcer in advanced pelvic organ prolapse: a case series. Int Urogynecol J. 2016 Jul;27(7):1057-62. doi: 10.1007/s00192-015-2930-3. Epub 2015 Dec 30. PMID 26718780
- [Background] Thiagamoorthy G, Khalil A, Cardozo L, Srikrishna S, Leslie G, Robinson D. The value of vaginal packing in pelvic floor surgery: a randomised double-blind study. Int Urogynecol J. 2014 May;25(5):585-91. doi: 10.1007/s00192-013-2264-y. Epub 2013 Dec 6. PMID 24310987
- [Background] Westermann LB, Crisp CC, Oakley SH, Mazloomdoost D, Kleeman SD, Benbouajili JM, Ghodsi V, Pauls RN. To Pack or Not to Pack? A Randomized Trial of Vaginal Packing After Vaginal Reconstructive Surgery. Female Pelvic Med Reconstr Surg. 2016 Mar-Apr;22(2):111-7. doi: 10.1097/SPV.0000000000000238. PMID 26825408
- [Background] Mercier RJ, Zerden ML. Intrauterine anesthesia for gynecologic procedures: a systematic review. Obstet Gynecol. 2012 Sep;120(3):669-77. doi: 10.1097/AOG.0b013e3182639ab5. PMID 22914480
- [Background] Simavli S, Kaygusuz I, Kinay T, Akinci Baylan A, Kafali H. Bupivacaine-soaked absorbable gelatin sponges in caesarean section wounds: effect on postoperative pain, analgesic requirement and haemodynamic profile. Int J Obstet Anesth. 2014 Nov;23(4):302-8. doi: 10.1016/j.ijoa.2014.07.004. Epub 2014 Jul 18. PMID 25281438
- [Background] Haytoglu S, Kuran G, Muluk NB, Arikan OK. Different anesthetic agents-soaked sinus packings on pain management after functional endoscopic sinus surgery: which is the most effective? Eur Arch Otorhinolaryngol. 2016 Jul;273(7):1769-77. doi: 10.1007/s00405-015-3807-2. Epub 2015 Oct 28. PMID 26511988
- [Background] Buchanan MA, Dunn GR, Macdougall GM. A prospective double-blind randomized controlled trial of the effect of topical bupivacaine on post-operative pain in bilateral nasal surgery with bilateral nasal packs inserted. J Laryngol Otol. 2005 Apr;119(4):284-8. doi: 10.1258/0022215054020322. PMID 15949082
- [Background] Karaman E, Gungor G, Alimoglu Y, Kilic E, Tarakci E, Bozkurt P, Enver O. The effect of lidocaine, bupivacaine and ropivacaine in nasal packs on pain and hemorrhage after septoplasty. Eur Arch Otorhinolaryngol. 2011 May;268(5):685-9. doi: 10.1007/s00405-010-1432-7. Epub 2010 Dec 1. PMID 21120661
- Available data/document: Study Protocol — https://www.scribd.com/document/344597619/Study-Protocol
- Available data/document: Informed Consent Form — https://www.scribd.com/document/344597523/Consent-Form
- Available data/document: Individual Participant Data Set — https://www.scribd.com/document/344597573/Data-Collection-Spreadsheet
- Available data/document: Participant Documents — https://www.scribd.com/document/344597424/Participant-Documents